CLINICAL TRIAL: NCT01680601
Title: Effect of Remote Ischaemic Preconditioning in Cardiac Dysfunction and End-organ Injury Following Cardiac Surgery With Cardiopulmonary Bypass in Children.
Brief Title: Remote Ischaemic Preconditioning in Children Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Principal Investigator, Maribel Verdesoto, PhD student, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: GN12KH253
Record Dates: First submitted 2012-08-29; First posted 2012-09-07 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Ischaemic Reperfusion Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIPC group (Experimental): Patients assigned to this arm will go through a remote ischaemic preconditioning (RIPC)protocol
  Interventions: Procedure: Remote ischaemic preconditioning (RIPC)
- Control (Placebo Comparator): Patients assigned to this arm will not receive the intervention, however the protocol will be applied to a wooden block in order to maintain blinding to relatives and investigators.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Remote ischaemic preconditioning (RIPC) — RIPC will be performed by 3 cycles of 5 minute leg ischaemia induced by inflation of a blood pressure cuff to 40 mmHg above the patient's systolic pressure. This protocol will be performed at two phases: 24 hours before surgery and during anaesthesia immediately prior to surgery.
  Arms: RIPC group
Procedure: Placebo
  Arms: Control

SUMMARY:
Surgical correction of congenital heart defects in children requires the utilization of cardiopulmonary bypass, a technique that temporarily substitutes heart and lung functions during surgery. During this process the patient´s circulation is controlled by a bypass machine which provides several functions:

1. Controls the patient's blood flow by pumping of blood in the patient's body.
2. Controls the correct oxygen levels in the patient's blood.
3. Regulates the temperature and fluid level of the blood. This process triggers negative responses in the heart and throughout the whole body, potentially resulting in injury to the heart and other organs such as brain, kidneys and lungs.

Remote ischaemic preconditioning (RIPC) describes a procedure that could potentially reduce the injury to heart muscle during cardiac surgery. The procedure consists of the inflation of a blood pressure cuff on the child's leg for three 5 minute cycles. This process acts by briefly reducing blood flow to the leg muscle, which will then activate the body´s own protective mechanisms and thereby reduce heart injury.

Several animal studies have been used to help the understanding of the mechanisms behind this process, and trials in human adults have showed optimistic results; however evidence regarding the paediatric population is limited and necessary since children present different basal profiles, risks and requirements.

The investigators propose a randomized clinical trial assessing the efficacy of RIPC to provide protection against injury to the heart and other organs in children going through cardiac surgery using CPB at the Royal Hospital for Sick Children. The research project will have a translational approach, integrating basic molecular mechanisms to clinical outcome. The investigators hope it will allow the understanding and utilisation of the patient´s own protective mechanisms, reducing CPB-related injury and ultimately improving patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing cardiac surgery for correction of congenital heart defects utilizing cardiopulmonary bypass and cold blood cardioplegia strategy of myocardial protection.
* Children whose parents understand the child's condition, the purpose of the study and are willing to participate.

Exclusion Criteria:

* Children whose parents either are unwilling or do not have sufficient understanding of the study.
* Emergency operations, where there is insufficient time to establish the study protocol.
* Premature children presenting a corrected gestational age under 35 weeks.
* Presence of extracardiac abnormalities, apart from cases of Down and DiGeorge syndromes which will be included.
* Patients with known viral blood infections (e.g. HIV, Hepatitis B) or severe congenital infection.
* Patients with severe preoperative brain injury.

Ages: 2 Days to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Measurement of the final cardiac injury after cardiopulmonary bypass assessed by markers of cardiac injury and echocardiography. | Pre and post operatively (immediately before and after surgery, 24 and 48 hours after surgery)
  Echocardiography assessment will take place before surgery, 24 and 48 hours after surgery. Blood markers of cardiac injury: B-type natriuretic peptide and Troponin will be measured before surgery, immediately after surgery, 24 and 48 hours after surgery in order to establish changes in the markers between the mentioned pre and post-operative time points.

SECONDARY OUTCOMES:
Protein and mRNA expression in the cardiac tissue related to the preconditioning process. | Expression assessed at the time of tissue extraction
  Cardiac tissue will be obtained only from patients who require tissue excision as part of the surgical procedure. Protein and mRNA expression will be assessed after extraction.
End organ damage assessment by measurement of markers relevant to lung and kidney function and evaluate a possible benefit from preconditioning. | Pre and post operatively (immediately before and after surgery, 24 and 48 hours after surgery)
  Blood markers (creatinin, cystatin C, Neutrophil gelatinase associated lipocalin,cGMP and Phosphodiesterase 5)will be measured before surgery, immediately after surgery, 24 and 48 hours after surgery in order to establish changes in the markers between the mentioned pre and post-operative time points.
Systemic immune response assessment by measurement of inflammatory mediators such as cytokines and nitric oxide metabolites. | Pre and postoperatively (immediately before and after surgery, 24 and 48 hours after surgery)
  Inflammatory blood markers (MDA, isoprostanes, NO metabolites, Cytokines, adhesion molecules, among others)will be measured before surgery, immediately after surgery, 24 and 48 hours after surgery in order to establish changes in the markers between the mentioned pre and post-operative time points

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hospital for Sick Children - Yorkhill, Glasgow, United Kingdom